CLINICAL TRIAL: NCT02108197
Title: Obstructive Sleep Apnea and Gestational Diabetes : Incidence and Effects of Continuous Positive Airway Pressure Treatment on Glucose Metabolism
Brief Title: Sleep Apnea and Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Sirimon Reutrakul, Associate Professor of Medicine, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-56-39
Record Dates: First submitted 2014-03-17; First posted 2014-04-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Gestational Diabetes; Sleep Apnea
MeSH Terms: conditions — Diabetes, Gestational; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP Intervention (Experimental): Continuous positive airway pressure (S9, ResMed)
  Interventions: Device: Continuous positive airway pressure (S9, ResMed)
- Wait-list (No Intervention): Wait list controls

INTERVENTIONS:
Device: Continuous positive airway pressure (S9, ResMed)
  Arms: CPAP Intervention

SUMMARY:
The investigators hypothesize that pregnant women with gestational diabetes will have a high incidence of sleep apnea, and that the treatment of sleep apnea will lead to improved glucose control in these women.

ELIGIBILITY:
Inclusion Criteria:

* gestational diabetes

Exclusion Criteria:

* pre-gestational diabetes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | two weeks
  Measuring glucose, fructosamine and insulin levels following a mixed meal test at 0 and 2 weeks. Glucose and insulin will be measured at 0 minutes and every 30 minutes thereafter for 2 hours. Fructosamine will be measured at 0 minutes only.

CONTACTS AND LOCATIONS:
Overall Officials: Sirimon Reutrakul, MD, Principal Investigator — Faculty of Medicine Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Chirakalwasan N, Amnakkittikul S, Wanitcharoenkul E, Charoensri S, Saetung S, Chanprasertyothin S, Chailurkit LO, Panburana P, Bumrungphuet S, Thakkinstian A, Reutrakul S. Continuous Positive Airway Pressure Therapy in Gestational Diabetes With Obstructive Sleep Apnea: A Randomized Controlled Trial. J Clin Sleep Med. 2018 Mar 15;14(3):327-336. doi: 10.5664/jcsm.6972. PMID 29458699